CLINICAL TRIAL: NCT03100253
Title: Open-label, Randomized Controlled Trial Comparing Tocilizumab to Anti-TNF Treatment and Discovery of Biomarkers for Treatment Selection in Rheumatoid Arthritis Patients With Inadequate Response to a First Anti-TNF
Brief Title: Rheumatoid Arthritis Treatment After First Anti-TNF INvestiGation
Acronym: RAFTING
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recrutiment
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRFMN-RA-6453
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Tocilizumab; anti-TNF treatment
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Etanercept; Infliximab; Adalimumab; golimumab; Certolizumab Pegol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Switching" strategy (Experimental): Tocilizumab [RoActemra®] [ATC: L04AC07] 8 mg/kg i.v. every 4 weeks OR 162 mg s.c every seven days
  Interventions: Drug: Tocilizumab
- "Cycling" strategy (Active Comparator): 1. Etanercept if initial failure to monoclonal antibodies: infliximab, adalimumab, golimumab or certolizumab OR
  2. Infliximab, adalimumab, golimumab or certolizumab if initial failure to the receptor fusion protein, etanercept.
  Interventions: Drug: Etanercept; Drug: Infliximab; Drug: Adalimumab; Drug: Golimumab; Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Tocilizumab — 8 mg/kg i.v. every 4 weeks OR 162 mg s.c every seven days
  Arms: "Switching" strategy
Drug: Etanercept — a. Etanercept if initial failure to monoclonal antibodies: infliximab, adalimumab, golimumab or certolizumab
  Arms: "Cycling" strategy
Drug: Infliximab — infliximab if initial failure to the receptor fusion protein, etanercept.
  Arms: "Cycling" strategy
Drug: Adalimumab — adalimumab if initial failure to the receptor fusion protein, etanercept.
  Arms: "Cycling" strategy
Drug: Golimumab — golimumab if initial failure to the receptor fusion protein, etanercept.
  Arms: "Cycling" strategy
Drug: Certolizumab Pegol — Certolizumab Pegol if initial failure to the receptor fusion protein, etanercept.
  Arms: "Cycling" strategy

SUMMARY:
To compare the efficacy of switching to a different molecular target (from TNF to IL6) versus cycling to a second TNF inhibitor in patients with active RA, who have not adequately responded to a previous treatment with a first anti-TNF.

DETAILED DESCRIPTION:
New drugs for the treatment of rheumatoid arthritis (RA) with action on specific molecular target (e.g. anti-TNF) have improved the prognosis of patients with an inadequate response to conventional therapy such as methotrexate (MTX).

However, approximately 50% of patients treated with first-line anti-TNF discontinue treatment after two years due to ineffectiveness or adverse events. The second line treatment involves the use of another anti-TNF drug or switching to a different molecular target (anti-IL6, -CD20 or CTLA-4-Ig) in combination with MTX.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent form and either male or female.
* Diagnosis of RA according to the 1987 ACR classification criteria OR 2010 ACR/EULAR classification criteria at least 6 months prior to screening.
* Patients with persistent RA disease activity whilst being treated with an initial TNFi agent on a background MTX up to 20-25 mg/week for at least 12 weeks defined according to SIR and EULAR guidelines as: primary non-response: failing to improve DAS28 by ≥ 1.2 or failing to achieve DAS28 ≤ 3.2 within the first three to six months of starting the initial TNFi; secondary non-response: determined by physician decision with evidence of flare and deterioration in DAS28 of ≥ 1.2.
* Methotrexate (MTX) dose stable for 28 days prior to screening.
* Patients on NSAIDs and / or corticosteroids must remain on an unchanged regimen for at least 28 days prior to study drug administration.
* The patient must be able to comply with the study visit schedule and other protocol requirements.
* The patient understands the purpose of the study and is able and willing to sign the informed consent form, according to ICH/GCP.
* Signed written informed consent for biological analysis.
* Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to start of trial. Women of childbearing potential and male patients must be willing to practice acceptable methods of contraception during treatment and for 6 months (female patients) and 3 months (male patients) after discontinuation of treatment.

Exclusion Criteria:

* Patients who have previously received more than 1 TNFi drug OR any other biological therapy.
* Patients with inflammatory joint disease of different origin or any arthritis with onset prior to 16 years of age.
* Patients taking any disease-modifying antirheumatic drug (DMARDs) (e.g. all except methotrexate). Discontinuation must occur at least 28 days prior to study treatment start.
* History or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug.
* Known hypersensitivity to any active substance or excipients of study drug.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with good EULAR | 24 weeks
  the proportion of patients with good EULAR response

SECONDARY OUTCOMES:
Proportion of patients with a good/moderate EULAR | 12 weeks
  Proportion of patients with a good/moderate EULAR response
Proportion of patients with a good/moderate EULAR | 24 weeks
  Proportion of patients with a good/moderate EULAR response
Proportion of patients with ACR20/50/70 response | 12 weeks
  Proportion of patients with ACR20/50/70 response
Proportion of patients with ACR20/50/70 response | 24 weeks
  Proportion of patients with ACR20/50/70 response
Proportion of patients with a remission according to DAS28/SDAI/CDAI | 24 weeks
  Proportion of patients with a remission according to DAS28/SDAI/CDAI
Proportion of patients with a remission according to DAS28/SDAI/CDAI | 48 weeks
  Proportion of patients with a remission according to DAS28/SDAI/CDAI
Proportion of patients with a remission according to DAS28/SDAI/CDAI | 96 weeks
  Proportion of patients with a remission according to DAS28/SDAI/CDAI
Van Der Heijde Modified Total Sharp Score [X-ray score] | 48 weeks
  Van Der Heijde Modified Total Sharp Score [X-ray score]
Van Der Heijde Modified Total Sharp Score [X-ray score] | 96 weeks
  Van Der Heijde Modified Total Sharp Score [X-ray score]
Health Assessment Questionnaire (HAQ) score | 24 weeks
  Health Assessment Questionnaire (HAQ) score
Health Assessment Questionnaire (HAQ) score | 48 weeks
  Health Assessment Questionnaire (HAQ) score
Health Assessment Questionnaire (HAQ) score | 96 weeks
  Health Assessment Questionnaire (HAQ) score

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Galeazzi, Principal Investigator — Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria alle Scotte
Locations (22):
- Italy (22):
  - Azienda Consorziale Ospedaliera Policlinico, Bari
  - Azienda Socio Sanitaria Territoriale - Papa Giovanni XXIII, Bergamo
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Ospedale Centrale di Bolzano, Bolzano
  - Azienda Ospedaliera Universitaria Policlinico Vittorio Emanuele, Catania
  - Azienda Ospedaliera-Universitaria S.Anna c/o Nuovo Arcispedale S. Anna, Cona
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo
  - Università di Firenze, Florence
  - Azienda Ospedaliera Universitaria Di Messina, Messina
  - Istituto Ortopedico Gaetano Pini, Milan
  - Azienda Ospedaliera Universitaria Policlinico di Modena, Modena
  - Policlinico Universitario Monserrato, Monserrato
  - Asl Napoli 1 centro, Napoli
  - Ospedale Maggiore di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale SS Annunziata, Sassari
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza, Torino
  - Ospedale Santa Chiara, Trento
  - Azienda Sanitaria Universitaria Integrata di Udine Sanata Maria della Misericordia, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona - Policlinico GB Rossi, Verona

IPD SHARING:
Plan to Share IPD: Undecided